CLINICAL TRIAL: NCT01779557
Title: The Prospective, Randomized, Parallel, Controlled, Multi-center Clinical Study of Huaren Peritoneal Dialysate and Baxter Peritoneal Dialysate
Brief Title: Safety and Effectiveness Evaluation of Two Kinds of Peritoneal Dialysate
Acronym: SEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Professor, Chief physician, Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-PD-2012; ChiCTR-TRC-13003001 (Registry Identifier: Chinese Clinial Trial Registry)
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Kidney Failure,Chronic
Keywords: CAPD; efficacy; safety; survival rate
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huaren peritoneal dialysate (Experimental): Huaren Peritoneal dialysate CAPD 3-5 times/d
  Interventions: Drug: Huaren Peritoneal Dialysate
- Baxter Peritoneal Dialysate (Active Comparator): Baxter Peritoneal dialysate CAPD 3-5 times/d
  Interventions: Drug: Baxter Peritoneal Dialysate

INTERVENTIONS:
Drug: Huaren Peritoneal Dialysate — Huaren Peritoneal dialysate CAPD 3-5 times/d
  Arms: Huaren peritoneal dialysate
Drug: Baxter Peritoneal Dialysate — Baxter Peritoneal dialysate CAPD 3-5 times/d
  Arms: Baxter Peritoneal Dialysate

SUMMARY:
This study is to evaluate the effectiveness and safety of Huaren Peritoneal Dialysate and Baxter Peritoneal Dialysate, investigate the proper dialysis dose for Chinese CAPD patients.

DETAILED DESCRIPTION:
This study is a prospective, randomized, parallel, controlled, multi-center clinical study of Huaren Peritoneal Dialysate and Baxter Peritoneal Dialysate.It aims to investigate the proper dialysis dose for Chinese CAPD patients.At the same time,it can evaluate the effectiveness and safety of Chinese product Huaren Peritoneal Dialysate and peritoneal dialysis product Baxter Peritoneal Dialysate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, male or female
* Patients with end stage renal diseases
* Dialysis mode: CAPD
* Dialysis duration:≥30 days and ≤6 months
* Be capable of implementing home dialysis
* Diabetic nephropathy, 3ml/min≤ residual renal GFR ≤15ml/min; other renal diseases, 3ml/min≤ residual renal GFR ≤10ml/min
* Sign the written informed consent

Exclusion Criteria:

* Acute renal failure
* Planing to receive kidney transplantation in 2 years
* Hemodialysis
* Exit site infection or tunnel infection
* Presenting 2/3 of the following: a. abdominal pain, turbid ascites, with or without fever; b. drainage fluid WBC>100×106/L, neutrophil ratio>50%; c.culture positive/ Gram stain positive in drainage fluid;
* Anti-HIV positive
* Allergic to components of dialysate
* Active, residual malignant tumor, or systemic infection, liver cirrhosis, severe congestive heart failure, anemia（Hb<80g/L）,malnutrition（Serum Alb<28g/L）,refractory hypertension
* Identified peritoneal high transportation by peritoneal equilibration test (PET)
* Extreme body shape (height> 185cm or height <145cm), obesity (BMI ≥ 33kg/m2)
* Poor compliance
* Pregnant or lactating, women of childbearing age do not agree to use effective contraceptive measures during the trial
* Has a history of alcoholism and drug abuse (defined as illegal drugs)
* Any circumstances when patients are believed unsuitable for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
survival rate | 1,2,3,4,5 years

SECONDARY OUTCOMES:
PD technique survival rate | 1,2,3,4,5 years
estimated glomerular filtration rate decline | 1,2,3,4,5 years
nutritional status | 1,2,3,4,5 years
quality of life(SF-36) | 1,2,3,4,5 years
cardiovascular events | 1,2,3,4,5 years
increments of dialysis dose | 1,2,3,4,5 years
medical costs | 1,2,3,4,5 years
dropout rate | 1,2,3,4,5 years

OTHER OUTCOMES:
AE, vital signs, laboratory tests | 1,2,3,4,5 years
peritonitis | 1,2,3,4,5 years
quality of products | 1,2,3,4,5 years
allergy to PD fluids, bags and tubes | 1,2,3,4,5 years

CONTACTS AND LOCATIONS:
Overall Officials: CHEN Xiangmei, yes, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou J, Cao X, Lin H, Ni Z, He Y, Chen M, Zheng H, Chen X. Safety and effectiveness evaluation of a domestic peritoneal dialysis fluid packed in non-PVC bags: study protocol for a randomized controlled trial. Trials. 2015 Dec 29;16:592. doi: 10.1186/s13063-015-1131-1. PMID 26715594